CLINICAL TRIAL: NCT02665923
Title: Gastric Emptying in Pediatric Patients
Brief Title: Gastric Emptying in Neonates and Infants After Formula Feeding
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Lena S. Sun, Emanuel M. Papper Professor of Anesthesiology and Professor of Pediatrics, Columbia University
Other Study IDs: AAAP6304
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Gastric Emptying

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Newborn (gastric emptying): A total of 100 healthy newborns who will be given formula feeding of known volume, and then serial ultrasound imaging of gastric antral volume will be performed until gastric emptying. Follow up of these newborns at two later time intervals will be performed (between ages 4-6 months, and 9-12 months).
  Interventions: Other: Gastric ultrasound
- Infants (4-6mons): 50 Patients will undergowill be given formula feeding of known volume, and then serial ultrasound imaging of gastric antral volume will be performed until gastric emptying.
- Infants (9-12 months): 50 Patients will undergowill be given formula feeding of known volume, and then serial ultrasound imaging of gastric antral volume will be performed until gastric emptying.

INTERVENTIONS:
Other: Gastric ultrasound — Ultrasound of abdomen to assess antral volume
  Groups: Newborn (gastric emptying)

SUMMARY:
Ultrasound imaging will be used to evaluate time for gastric emptying in healthy, fasting newborns, and infants following feeding of clear liquids and/or milk (including breast or formula).

DETAILED DESCRIPTION:
The study involves serial ultrasounds over several visits. Healthy newborns in the Newborn Nursery will be recruited to conduct this study. The study will include a total of 50 healthy newborns who will be given formula feeding of known volume, and then serial ultrasound imaging of gastric antral volume will be performed until gastric emptying.

The study originally was designed to perform follow up of these newborns at two later time intervals (between ages 4-6 months, and 9-12 months). The purpose of follow-up is to evaluate whether there are age-related changes in gastric emptying. Due to the pause/suspension of research activity during the pandemic, these follow up studies of the original newborn cohort could not be completed. The protocol is thus revised as follows:

The study will recruit 50 4-6 months old and 50 9-12months old infants and perform gastric emptying serial ultrasound to evaluate if there are age-related changes in gastric emptying.

ELIGIBILITY:
Inclusion criteria for study cohort are pediatric patients from Allen Hospital and Morgan Stanley Children's Hospital of New York Presbyterian Hospital who are receiving feeding by formula

1. healthy full-term (postmenstrual age ≥ 36 weeks) newborns aged 0-5 days or
2. healthy infants (4-6 months old and 9-12 months old)

Exclusion criteria are individuals who have

1. newborn history of requirement resuscitation at delivery
2. newborn history of admission to the Neonatal Intensive Care Unit
3. any history of hospital admission
4. history of gastroesophageal reflux or other feeding difficulty
5. receiving any medication known to accelerate or delay gastric emptying, including but not limited to opioid-containing medications and antacids.

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will be performing serial ultrasounds in total of 100 healthy newborns, and 50 4-6 months old and 50 9-12 months old infants.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2016-03; Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Gastric Antral Volumes in Newborns | Up to 6 hours
  To determine gastric emptying time in newborns, serial gastric antral volumes will be measured before and after formula feeding until return to baseline measurements at 10-15 minute intervals.

SECONDARY OUTCOMES:
Gastric Antral Volumes in Infants | Up to 6 hours
  To determine gastric emptying time in 4-6 months old and 9-12 months old infants. serial gastric antral volumes will be measured before and after formula feeding until return to baseline measurements at 10-15 minute intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Lena S. Sun, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center / NewYork-Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Sharing through written communication and request to PI
Supporting Information: Study Protocol
Time Frame: Available within 12 months after analysis of results is completed and published.
Access Criteria: Upon review and request.